CLINICAL TRIAL: NCT06862089
Title: A Prospective Study Evaluating the Impact of Conservative Management on Retained Products of Conception and EMV
Status: Recruiting | Type: Observational
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Huang Rui, MD,Gynecologist, Department of Hysteroscopy Center, Fu Xing Hospital, Capital Medical University
Other Study IDs: 2024FXHEC-KSP073
Record Dates: First submitted 2025-02-12; First posted 2025-03-06 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Retained Products of Conception; Miscarriage; Conservative Management
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the therapeutic effects of the conservative treatment approach on pepole with retained products of conception (RPOC) and Enhanced myometrial vascularity (EMV).

The main question it aims to answer is: Is it possible to achieve the natural resolution of RPOC by combining it with EMV through conservative treatment？ Participants will receive conservative treatment (such as mifepristone, GnRH-a, or expectant management) following the initial diagnosis of RPOC and EMV, and the therapeutic efficacy of the conservative approach will be assessed after the completion of two menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

* Recent history of miscarriage or delivery (within the past 8 weeks)
* Strong willingness to undergo conservative management
* Hemodynamically stable
* Signed informed consent form

Exclusion Criteria:

* Heavy vaginal bleeding (requiring immediate surgical intervention)
* Active pelvic or systemic infection (e.g., fever >38°C, elevated CRP/WBC)
* Severe dysfunction of vital organs (heart, liver, or kidney)
* Known drug allergies or contraindications to proposed medications (e.g., misoprostol intolerance)
* Suspected ectopic pregnancy or gestational trophoblastic disease (confirmed by ultrasound or β-hCG levels)
* Placenta accreta spectrum disorders diagnosed during current pregnancy
* History of uterine artery embolization

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population of who visited the outpatient department of the hysteroscopy center of our hospital from October 2024 to October 2026 and were provisionally diagnosed as " retained products of conception (RPOC)" based on their history and symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The disappearance rate of RPOC | After conservative treatment, transvaginal ultrasound was performed at the end of the second menstrual cycle (calculated from the first day of menses, 28-30 days per cycle) to assess RPOC resolution
  The definition of "the disappearance rate of RPOC" refers to the absence of significant residual trophoblastic tissue as indicated by ultrasound examination

SECONDARY OUTCOMES:
the disappearance rate of EMV | Immediately after the completion of conservative treatment
  The definition of "the disappearance rate of EMV" refers to a PSV (Peak Systolic Velocity) of less than 20 cm/s or its complete disappearance as indicated by Ultrasound Doppler examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Hysteroscopy Center, Fuxing Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication